CLINICAL TRIAL: NCT05133388
Title: The Prevelence of HBB c.93-21 G-A Gene Mutation in Suspected Cases of β Thalassemia in Assiut University Hospitals.
Brief Title: The Prevelence of HBB c.93-21 G-A in β Thalassemia Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Amira Saber Hamed Ahmed, ASHAhmed, Assiut University
Other Study IDs: β thalassemia gene mutation
Record Dates: First submitted 2021-11-03; First posted 2021-11-24 (Actual); Last update posted 2023-01-31 (Actual); Status verified 2023-01

CONDITIONS: Beta-Thalassemia
MeSH Terms: conditions — beta-Thalassemia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Genetic: ARMS PCR — ARMS PCR using primer pairs that only amplify individual alleles

SUMMARY:
* To design an amplification-refractory mutation system (ARMS) for the DNA diagnosis of the IVS I-110 (G>A) [HBB:c.93-21G˃A] mutation.
* To detect the prevelence of the mutation among Assiut University Hospital patients.
* Phenotype/genotype correlation of the mutation.

DETAILED DESCRIPTION:
* The β-thalassaemias result from over 300 gene mutations (Kurtoğlu A,et al 2016)
* These mutations are regionally specific and the spectrum of mutations has been determined for most at-risk populations. The strategy for identifying β-thalassaemia mutations is usually based on knowledge of the common mutations in the ethnic group of the individual being screened (Old JM, 2007).

The β globin gene mutation [HBB:c.93-21G˃A] or IVS I-110 (G>A) is the most common β globin gene mutation in the Mediterranean region (Old JM, 2007). . There is no consensus about the % of the mutation among β thalassemic patients in Egypt [has been reported (25.8%) by El-Gawhary et al. 2007, (33.75%) by Soliman et al. 2010, (48%) by El-Shanshory et al. 2014, (22%) by Elmezayen et al. 2015 and (34%) by Elhalfawy et al. 2017].

According to the HbVar site, it represents 33% of the β globin gene mutations in the Egyptians. 28.5% according to Henderson S ,et al 2009 .

* The mechanism of this mutation depends on formation of a new splicing site resulting in 80% abnormal spliced mRNA and 20% normal mRNA .
* The molecular characterization of the globin gene mutation is necessary for definite diagnosis, genetic counseling, and in prenatal diagnosis.
* The amplification-refractory mutation system (ARMS) is a simple method for detecting any mutation involving single base changes or small deletions.
* The DNA is analyzed after amplification by PCR for Detection of point mutation IVS I-110 (G>A) by Using primer pairs that only amplify individual alleles.

ELIGIBILITY:
Inclusion Criteria:

* β thalassemia (suspected & clinically diagnosed cases)

Exclusion Criteria:

* Iron deficiency anaemia, anaemia of chronic disease, types of haemolytic anaemias other than thalassemia, other types of thalassemia and Hb variants.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Assiut University Hospitals patients
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2023-01-30 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Introduction of arms pcr in diagnosis . | 2 years
  To introduce the ARMS PCR as a cheap and simple DNA diagnostic tool for any point mutation
Database initation . | 2 years
  Initiating database of haemoglobinopathesis by registering data.

CONTACTS AND LOCATIONS:
Overall Officials: Ola Afifi, Study Director — Assiut University
Locations (1):
- Faculty of Medicine Assiut University, Asyut, Egypt

REFERENCES:
- [Background] Henderson S, Timbs A, McCarthy J, Gallienne A, Van Mourik M, Masters G, May A, Khalil MS, Schuh A, Old J. Incidence of haemoglobinopathies in various populations - the impact of immigration. Clin Biochem. 2009 Dec;42(18):1745-56. doi: 10.1016/j.clinbiochem.2009.05.012. Epub 2009 Jun 1. PMID 19497317
- [Background] Old JM. Screening and genetic diagnosis of haemoglobinopathies. Scand J Clin Lab Invest. 2007;67(1):71-86. doi: 10.1080/00365510601046466. PMID 17365985
- [Background] El-Gawhary S, El-Shafie S, Niazi M, Aziz M, El-Beshlawy A. Study of beta-Thalassemia mutations using the polymerase chain reaction-amplification refractory mutation system and direct DNA sequencing techniques in a group of Egyptian Thalassemia patients. Hemoglobin. 2007;31(1):63-9. doi: 10.1080/03630260601057104. PMID 17365006
- [Background] Soliman OE, Yahia S, Shouma A, Shafiek HK, Fouda AE, Azzam H, Abousamra NK, Mahfouz R, Goda EF, El-Sharawy SA. Reverse hybridization StripAssay detection of beta-thalassemia mutations in northeast Egypt. Hematology. 2010 Jun;15(3):182-6. doi: 10.1179/102453310X12583347010214. PMID 20557680
- [Background] El-Shanshory M, Hagag A, Shebl S, Badria I, Abd Elhameed A, Abd El-Bar E, Al-Tonbary Y, Mansour A, Hassab H, Hamdy M, Alfy M, Sherief L, Sharaf E. Spectrum of Beta Globin Gene Mutations in Egyptian Children with beta-Thalassemia. Mediterr J Hematol Infect Dis. 2014 Nov 1;6(1):e2014071. doi: 10.4084/MJHID.2014.071. eCollection 2014. PMID 25408857
- [Background] Elmezayen AD, Kotb SM, Sadek NA, Abdalla EM. beta-Globin Mutations in Egyptian Patients With beta-Thalassemia. Lab Med. 2015 Winter;46(1):8-13. doi: 10.1309/LM1AYKG6VE8MLPHG. PMID 25617386
- [Background] Kurtoglu A, Karakus V, Erkal O, Kurtoglu E. beta-Thalassemia gene mutations in Antalya, Turkey: results from a single centre study. Hemoglobin. 2016 Nov;40(6):392-395. doi: 10.1080/03630269.2016.1256818. Epub 2017 Mar 3. PMID 28276871